CLINICAL TRIAL: NCT04071951
Title: A Multicenter RCT of Pharmacist-Directed Transitional Care to Reduce Post-Hospitalization Utilization
Brief Title: Pharmacist Intervention to Reduce Post-Hospitalization Utilization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Josh Pevnick, Associate Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00053414; R01AG058911 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Nonadherence, Patient; Polypharmacy; Readmission
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Arm (Experimental): Pharmacist-Led Medication Reconciliation, Regimen Review, and Adherence and Literacy Assessment and Counseling
  Interventions: Behavioral: Pharmacist-led Hospital Discharge Care Intervention
- Usual Care (No Intervention): Patients in this study will receive usual care. Clinically-indicated services, including pharmacist services, may be provided to control group patients.

INTERVENTIONS:
Behavioral: Pharmacist-led Hospital Discharge Care Intervention — Pharmacists will address medication reconciliation, medication adherence, and polypharmacy issues as appropriate. Pharmacists will rely most on their prior training, but study investigators will also encourage the use of documentation templates with reminders, Beers list, deprescribing, motivational interviewing, the Medication Adherence and Literacy tool, and post-discharge phone calls.
  Pharmacists will assess patient needs and customize accordingly. All patients will receive one discharge counseling visit and one post-discharge phone call, but pharmacists will find that some patients need further phone calls, interventions, referrals, or other interactions. Some or all of the pharmacist activities may take place over the phone.
  Arms: Pharmacist Arm

SUMMARY:
This is a randomized trial testing a peri- and post-discharge pharmacist-led medication management intervention on post-discharge utilization, including both readmissions and emergency department visits within 30 days of discharge. The intervention incorporates evidence addressing three main areas: medication reconciliation, medication adherence, and polypharmacy.

This study uses a pragmatic trial randomized at the patient level and conducted in two large hospitals to achieve the following aims, each of which has been designed using the RE-AIM framework:

Aim 1: To test the effect of PHARM-DC on post-discharge utilization among patients most at risk for post-discharge ADEs: recently discharged older adults taking >10 medications or >3 high-risk medications using a prospective, randomized, pragmatic multi-site study.

Aim 2: To study barriers and facilitators of implementing PHARM-DC using a qualitative study.

Aim 3: To analyze the costs of PHARM-DC, including the incremental cost per readmission averted and the net incremental cost from the health system perspective using a time-and-motion study and a cost-effectiveness analysis.

DETAILED DESCRIPTION:
There are three components to this study: (1) the prospective, randomized, controlled trial (RCT), which includes a pharmacist-led hospital discharge care intervention, (2) the qualitative study, which involves focus groups and interviews, and (3) a cost-effectiveness study, which involves a review of the literature and a time-and-motion study component.For all three studies, there are two sites: CSMC and Brigham and Women's Hospital in Boston. Additionally, Dr. Kennelty of University of Iowa will participate in the qualitative study.1. For the RCT: Eligible patients will be identified through the use of a daily Epic report using inclusion/exclusion criteria. Patients will be randomized by a study coordinator to the intervention arm or control arm. For the control arm, patients will receive usual care, which includes medication reconciliation at hospital admission. For the intervention arm, pharmacy staff will address medication reconciliation at hospital discharge, medication review, and medication adherence. Most intervention activities will occur during the hospital stay or during a post-discharge phone call. We estimate a total number of 4,888 patients per study arm.

2. For the qualitative study: This is a qualitative study employing focus groups aimed at understanding implementation barriers and facilitators. Dr. Kennelty and study staff will conduct 3-day site visits to hold focus groups and/or interviews regarding intervention expectations, how the intervention is being implemented, barriers/facilitators to adoption and implementation, and adaptations made during delivery. Towards the end of the trial, Dr. Kennelty and study staff will use phone interviews to determine any changes to the implementation of PHARM-DC that occurred during the RCT, as well as to understand whether and how institutions will address the maintenance of PHARM-DC after the study ends. We estimate that up to 180 people may participate in this qualitative study.

3. For the cost-effectiveness study: This is a time-and-motion study aimed at understanding how much time during the day pharmacists spend on activities related to the hospital discharge (and post-discharge) interventions. During the trial, we will use time and motion methodology to understand how much pharmacist time is needed for PHARM-DC. Coupled with data on post-discharge utilization, this will enable us to conduct economic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a medical ward, AND
* > 55 years AND
* ≥ 10 prescription medications at admission

OR

• ≥ 3 high-risk medications (anticoagulants, antiplatelets, insulin, oral hypoglycemics) at admission

Exclusion Criteria:

* Expected discharge to another state, acute care facility, psychiatric facility, or locked facility (including locked skilled nursing facility, jail, or prison) OR
* Expected AMA or left hospital against medical advice (AMA) OR
* Homeless OR
* On hospice OR
* Already enrolled into study within the past year OR
* Patients admitted by admitting or attending Primary Medical Doctors who have a specialty that is not Internal Medicine or Family Medicine OR
* Expected to receive pharmacist-led peri- and post-discharge medication management regardless of the trial OR
* Expected post-discharge setting not conducive to the studied medication management intervention (e.g. SNF, rehabilitation facility) OR
* Patients admitted with a suspected or confirmed diagnosis of COVID-19.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6478 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2026-01-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Pevnick, Principal Investigator — Associate Professor of Medicine
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murry LT, Keller MS, Pevnick JM, Schnipper JL, Kennelty KA; PHARM-DC Group. A qualitative dual-site analysis of the pharmacist discharge care (PHARM-DC) intervention using the CFIR framework. BMC Health Serv Res. 2022 Feb 12;22(1):186. doi: 10.1186/s12913-022-07583-5. PMID 35151310
- [Derived] Pevnick JM, Keller MS, Kennelty KA, Nuckols TK, Ko EM, Amer K, Anderson L, Armbruster C, Conti N, Fanikos J, Guan J, Knight E, Leang DW, Llamas-Sandoval R, Matta L, Moriarty D, Murry LT, Muske AM, Nguyen AT, Phung E, Rosen O, Rosen SL, Salandanan A, Shane R, Schnipper JL. The Pharmacist Discharge Care (PHARM-DC) study: A multicenter RCT of pharmacist-directed transitional care to reduce post-hospitalization utilization. Contemp Clin Trials. 2021 Jul;106:106419. doi: 10.1016/j.cct.2021.106419. Epub 2021 Apr 28. PMID 33932574

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacist Arm: Pharmacist-Led Medication Reconciliation, Regimen Review, and Adherence and Literacy Assessment and Counseling
  Pharmacist-led Hospital Discharge Care Intervention: Pharmacists will address medication reconciliation, medication adherence, and polypharmacy issues as appropriate. Pharmacists will rely most on their prior training, but study investigators will also encourage the use of documentation templates with reminders, Beers list, deprescribing, motivational interviewing, the Medication Adherence and Literacy tool, and post-discharge phone calls.
  Pharmacists will assess patient needs and customize accordingly. All patients will receive one discharge counseling visit and one post-discharge phone call, but pharmacists will find that some patients need further phone calls, interventions, referrals, or other interactions. Some or all of the pharmacist activities may take place over the phone.
Period: Overall Study
Arm/Group | Pharmacist Arm | Usual Care
Started | 3239 | 3239
Completed | 3213 | 3215
Not Completed | 26 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist Arm | Usual Care | Total
Number analyzed (Participants) | 3213 | 3215 | 6428
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (10.2) | 75.6 (10.2) | 75.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1586 | 1577 | 3163
  Male | 1627 | 1638 | 3265
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 8 | 14
  Asian | 139 | 118 | 257
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 479 | 475 | 954
  White | 2303 | 2367 | 4670
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 286 | 247 | 533
Study Site [Count of Participants; unit: Participants]
  Cedars-Sinai Medical Center | 1299 | 1300 | 2599
  Brigham and Women's Hospital | 1914 | 1915 | 3829

OUTCOME MEASURES:

1. Primary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Including Hospitals at Least Statewide)
Description: A patient is readmitted to a hospital (including observation) or has an ED visit within 30 days of discharge (including all hospitals at least statewide), excluding foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations
Time Frame: Hospitalization to a hospital or ED visit within 30 days of discharge (checking at least all same state facilities)
Population: note that to obtain outside hospital data, analysis was restricted to 4602 patients with fee-for-service Medicare (for whom all-hospital claims data was available)
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Arm | Usual Care
Number analyzed (Participants) | 2288 | 2314
Participants | 595 | 610

2. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital)
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge, excluding foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

3. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital) Stratified by Receipt of Different Intervention Components
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge. This outcome measure will analyze the outcome by whether patients received the intervention components (admission medication reconciliation, medication regimen review, actions to improve adherence, side effect management, drug level monitoring, discharge medication reconciliation, patient/caregiver education, motivational interviewing, post-discharge follow-up phone call, medication access, communication with PCP, communication with communication pharmacy, other). The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

4. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital) Stratified by Whether Patient Has a Diagnosis of Congestive Heart Failure at Admission
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by whether patient has a diagnosis of congestive heart failure at admission. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

5. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital), Stratified by Whether Patient Has Three or More High Risk Medications (Anticoagulants, Antiplatelets, Insulin, Oral Hypoglycemics) Prior to Admission
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by whether patient has three or more high risk medications (anticoagulants, antiplatelets, insulin, oral hypoglycemics) prior to admission. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

6. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital), Stratified by Whether Patient Has 10 or More Medications Prior to Admission
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by whether patient has 10 or more medications prior to admission. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

7. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital) Stratified by Study Site
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by study site. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

8. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital) Stratified by Patient Medication Adherence and Literacy
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by patient medication adherence and literacy (as assessed by study pharmacists, in addition to using limited English proficiency as a proxy for low medication literacy). The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

9. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospitalization and ED Visits (Same-hospital) Stratified by Quintiles of Patient Socioeconomic Status (Estimated Via Median Income of Home Census Tract)
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by patient socioeconomic status (estimated via median income of home census tract). The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

10. Secondary Outcome: Rate (%) of New BZR Discharge Prescriptions Among Patients Not Taking BZRs Prior to Admission
Description: A dichotomous variable for a new discharge prescription of BZRs among patients not taking BZRs prior to admission.
Time Frame: Patients not taking BZRs prior to admission
Reporting Status: Not Posted

11. Secondary Outcome: Rate (%) of Increased BZR Dose Prescription Among Patients Taking BZRs Prior to Admission
Description: A dichotomous variable for an increased dose prescription among patients taking BZRs prior to admission.
Time Frame: Patients taking BZRs prior to admission
Reporting Status: Not Posted

12. Secondary Outcome: Rate (%) of Post-hospitalization Fall-related Injuries as Healthcare Utilization (Hospitalization, ED Visits, Urgent Care Visits, or Office Visits)
Description: The investigators define post-hospitalization fall-related injuries as healthcare utilization (hospitalization, ED visits, urgent care visits, or office visits) due to fall-related injuries within 30 days of discharge of the index admission. The investigators will link Medicare claims data to trial data to track this outcome at the individual patient level.
Time Frame: Fall-related injuries within 30 days of discharge of the index admission
Reporting Status: Not Posted

13. Secondary Outcome: Rate of 30 Day Post-discharge Hospitalizations and ED Visits (Same Hospital) Stratified by Patient Age Groups
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified by patient age groups. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

14. Secondary Outcome: Rate of 30 Day Post-discharge Hospitalizations and ED Visits (Same Hospital) Stratified According to Time Periods That Had Changes in the Intervention and Control Arms
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge stratified according to time periods that had changes in the intervention and control arms. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

15. Secondary Outcome: Rate of 30 Day Post Hospitalization in ED Visits (Same Hospital) Restricted to Medication-related Utilization
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge restricted to medication-related utilization. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

16. Secondary Outcome: Rate of 7 Day Post-discharge Hospitalization Medication-related Post-discharge Utilization.
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 7 days of discharge by hospitalization medication-related post-discharge utilization. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 7 days of discharge
Reporting Status: Not Posted

17. Secondary Outcome: Rate (%) of 30-day Post-discharge Hospital Utilization With ED Visits, Observation Stays, and Inpatient Readmissions Counted Separately (Including Hospitals at Least Statewide).
Description: A patient is readmitted to a hospital under inpatient or observation status or has an ED visit within 30 days of discharge (including hospitals at least statewide). The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to a hospital or ED visit within 30 days of discharge (checking at least all same state facilities)
Reporting Status: Not Posted

18. Secondary Outcome: 30-day, All-cause Mortality After Hospital Discharge
Description: All-cause mortality rate and survival analysis through Day 30 after hospital discharge.
Time Frame: Death occurring within 30 days after hospital discharge
Reporting Status: Not Posted

19. Secondary Outcome: Rate (%) of 30 Day Post-discharge Hospitalizations and ED Visits (Same Hospital) Among Patients Who Were Enrolled and Received the Intervention, Compared to Patients Who Were Eligible Yet Not Enrolled During the Study Period.
Description: A patient is readmitted to the same hospital (including observation stays) or has an ED visit within 30 days of discharge. The investigators will exclude foreseen readmissions, which include: transplants, chemotherapy or radiotherapy, treatment follow-up, rehabilitation care, and planned operations.
Time Frame: Hospitalization to the same hospital or ED visit within 30 days of discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of randomization (near hospital admission) up to 90 days after hospital discharge
Arm/Group | Pharmacist Arm | Usual Care
All-Cause Mortality (participants affected / at risk) | 330/3239 | 334/3239
Serious Adverse Events (participants affected / at risk) | 1485/3239 | 1438/3239
Other Adverse Events (participants affected / at risk) | 0/3239 | 0/3239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacist Arm (N=3239) | Usual Care (N=3239)
90-day post-discharge utilization (General disorders) | 1155 | 1104
30-day post-discharge utilization (same hospital) (General disorders) | 662 | 666

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04071951/Prot_SAP_000.pdf